CLINICAL TRIAL: NCT00447863
Title: An Open-Label, Single-Dose, Randomized, 2-Period, Crossover, Bioequivalence Study to Compare Levonorgestrel 90 mg/Ethinyl Estradiol 20 mg in 2 Dosage Forms With Different Dissolution Characteristics in Healthy, Cycling Women
Brief Title: Study Evaluating the Bioequivalence of Levonorgestrel/Ethinyl Estradiol Combinations in Cycling Women
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 0858A2-109
Record Dates: First submitted 2007-03-13; First posted 2007-03-15 (Estimated); Last update posted 2021-08-20 (Actual); Status verified 2021-08

CONDITIONS: Contraception
MeSH Terms: interventions — Ethinyl Estradiol-Norgestrel Combination

INTERVENTIONS:
Drug: Levonorgestrel/Ethinyl Estradiol

SUMMARY:
Levonorgestrel/ethinyl estradiol (LNG/EE) is an investigational drug that is being developed as an oral contraceptive (birth control pill). The purpose of this trial is to compare different preparations of LNG/EE by assessing the way they are absorbed into the blood.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 to 35 years.
* Healthy as determined by the investigator on the basis of medical history and screening evaluations.
* Must have a history of normal menstrual cycles (24 to 34 days) for the 3-month period preceding entry into the study.

Exclusion Criteria:

* Any surgical or medical condition that may interfere with the absorption, distribution, metabolism, or excretion of the test article.
* Presence, history, or family history of thrombophlebitis, thrombosis, or thromboembolitic disorders, deep vein thrombosis, pulmonary embolism, or known coagulopathy.
* Bethesda system report of low-grade squamous intraepithelial lesion or greater for a cervical cytologic smear obtained within the last 3 months.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2007-08; Study Completion 2007-08

PRIMARY OUTCOMES:
To assess the bioequivalence of 2 batches of LNG/EE tablets with different dissolution characteristics

SECONDARY OUTCOMES:
To obtain additional safety and tolerability data concerning LNG/EE in healthy, cycling women

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer